CLINICAL TRIAL: NCT05392088
Title: Characterization and Prognostic Role of Myocardial Injury in Patients With COVID-19. The CardioCOVID Gemelli Study.
Acronym: CardioCOVID
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, IRCCS Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4923
Record Dates: First submitted 2022-05-24; First posted 2022-05-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Injury; COVID-19
Keywords: Myocardial Injury; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Miocardial injury: Patients hospitalized at Policlinico Universitario A. Gemelli IRCSS since March 1, 2021, with a diagnosis of SARS-CoV-2 infection (≥1 positive nasopharyngeal swab) and at least one value of high-sensitivity cardiac troponin I (hs-cTnI) >99th percentile upper reference limit measured during the index hospitalization.
  Interventions: Other: DATA EXTRACTION; Other: FOLLOW-UP
- No Miocardial injury: Patients hospitalized at Policlinico Universitario A. Gemelli IRCSS since March 1, 2021, with a diagnosis of SARS-CoV-2 infection (≥1 positive nasopharyngeal swab) and value of high-sensitivity cardiac troponin I (hs-cTnI) <99th percentile upper reference limit.
  Interventions: Other: DATA EXTRACTION; Other: FOLLOW-UP

INTERVENTIONS:
Other: DATA EXTRACTION — For all patients enrolled Data Mart COVID-19 developed within Generator Real World will be used to automatically extract both structured and unstructured data from hospital databases of patients infected from SARS-CoV-2.The specific data that which will be exploited are:
  * Demographics data;
  * Patient comorbidities, vital signs and symptoms at the time of admission;
  * Laboratory analysis;
  * In-hospital complications (e.g.: need for non-invasive or invasive ventilation, access to intensive care unit, length of hospitalization, use of glucocorticoids or antibiotics, death);
  * Blood gas exchange information;
  * Radiological reports;
  * Medications at the time of admission, during hospitalization and at the time of discharge;
  * Vaccination status.
Other: FOLLOW-UP — All patients will undergo a clinical follow-up by telephonic interview and/or clinical visit at 12 months from hospital discharge, during which the incidence of MACE, dysrhythmias, inflammatory heart disease and/or thrombotic disorders (both as incidence of the composite and as incidence of each individual components) in the past months will be investigated.

SUMMARY:
The present retrospective and prospective observational study aims at evaluate the clinical predictors of myocardial injury in patients hospitalized for COVID-19 infection since the introduction of vaccines that could allow the development of predictive models as well as help clinicians in the early assessment of the risk of myocardial injury and the prevention of the associated unfavourable outcomes.

Furthermore, this study will characterize the cardiovascular outcomes in the post-acute COVID-19 phase, and it will evaluate for the first time the long-term clinical outcomes of patients who experienced myocardial injury, possibly paving the way for the implementation of specific therapies aiming to reduce the cardiovascular risk and the long- term sequelae of COVID-19.

DETAILED DESCRIPTION:
Background:

Coronavirus disease-2019 (COVID-19) is a global pandemic caused by the novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that is resulting in substantial morbidity and mortality (1). Of interest, a significant proportion of patients presenting with COVID-19 infection and requiring hospitalization demonstrate biomarker evidence of myocardial injury (defined as elevation in circulating cardiac troponin levels), which has been shown to be associated with increased risk of in-hospital morbidity (i.e.: rate of non- invasive and invasive ventilation, access to intensive care unit, length of hospitalization, use of glucocorticoids or antibiotics) and mortality (2-6). The pathogenesis of myocardial injury in COVID-19 is still unclear, with proposed mechanisms that include cytokine-mediated damage, oxygen supply-demand imbalance, ischemic injury from microvascular thrombi formation and direct viral invasion of the myocardium (7-9). Notably, the clinical predictors of myocardial injury in COVID-19 infection are still unknown, and, therefore, there is lack of therapeutic opportunities to prevent or reduce myocardial injury and the related-unfavourable outcomes.

Moreover, the post-acute sequelae of COVID-19 could potentially involve the pulmonary and several extrapulmonary organs, including the cardiovascular system (10). A few studies <<to date have investigated cardiovascular outcomes in the post-acute phase of the COVID-19, and most with a short duration of follow-up and a narrow selection of cardiovascular outcomes (11-13). Therefore, a comprehensive assessment of post-acute COVID-19 sequelae on the cardiovascular system is still missing and, of interest, studies addressing the post-acute COVID-19 sequelae in patients who developed myocardial injury during COVID-19 infection are lacking (14).

Given these shortcomings in this evolving area of clinical research, a comprehensive characterization of myocardial injury in patients with COVID-19 infection and the identification of clinical predictors for its occurrence could allow the development of predictive models, thus helping clinicians in the disease phenotyping and the early assessment of the risk of unfavourable outcome and improving a fast determination of most appropriate treatments and clinical paths, efficient planning and use of clinical resources in terms of treatment type and units (such as intensive care or coronary intensive care). In addition, the identification of clinical predictors and/or protective factors for myocardial injury in COVID-19 infection may pave the way for the development of specific therapeutic strategies aiming to reduce the impact of myocardial injury on COVID-19-related morbidity and mortality. Finally, assessing the long-term cardiovascular impact of myocardial injury in COVID-19 infection could help clinicians in the prognostic stratification and the choice of therapeutic strategies in the post-acute COVID-19 phases, possibly identifying those patients that may need a more aggressive therapy and a closer follow-up.

OBJECTIVES

Primary objective To identify clinical predictors of myocardial injury in patients hospitalized for COVID-19 infection since the introduction of vaccines (i.e., March 1, 2021).

Secondary objectives

1. To evaluate if the presence of myocardial injury during the index hospitalization for COVID-19 is associated with a worse in-hospital clinical course in terms of in-hospital complications and need for aggressive therapies.
2. To evaluate if the presence of myocardial injury during the index hospitalization for COVID-19 predicts a worse clinical outcome in terms of major adverse cardiovascular events (MACE) (defined as the composite of cardiovascular death, ischemic heart disease [acute or chronic coronary syndromes], stroke/transient ischemic attack [TIA] and hospitalization for heart failure), dysrhythmias (defined as the composite of new-onset atrial fibrillation and/or ventricular arrhythmias), inflammatory heart disease (pericarditis and/or myocarditis) or thrombotic disorders (pulmonary embolism, deep vein or superficial vein thrombosis) at 12-months follow-up.

Methods:

Study design Retrospective and prospective observational study.

All consecutive patients hospitalized at Policlinico Universitario A. Gemelli IRCSS since March 1, 2021, with a diagnosis of SARS-CoV-2 infection (≥1 positive nasopharyngeal swab) and at least one value of high-sensitivity cardiac troponin I (hs-cTnI) measured during the index hospitalization will be enrolled. Given that the patients are unable to physically sign the informed consent form due to epidemiological reasons (contamination of papers by SARS-CoV-2), each patient will verbally declare the consent to "Consenso al trattamento dei dati personali e dei campioni biologici a scopo di ricerca - no profit", "modulo di dichiarazione della volontà espresso ai fini del consenso informato generale alle cure" and "modulo dossier sanitario - richiesta di oscuramento/deoscuramento di eventi/episodi" at the presence of at least two witnesses.

Inclusion criteria will include:

* Age ≥18 years;
* Overt COVID-19 infection (molecular nasopharyngeal swab positive for SARS-CoV-2 ≥1);
* Patient with at least a high sensitivity Troponin I measured during hospitalization course.
* Available data on vaccination.
* Verbal informed consent

Exclusion criteria will include:

* Age <18 years;
* Patient in whom at least one high sensitivity Troponin I value measured during the course of hospitalization is not available.
* No data available on vaccination status.

This study will make use of Data Mart COVID-19 developed within Generator Real World Data Unit. The Data Mart COVID-19 belongs to the family of the diagnostic and prognostic mini-bots developed within the Generator Real World Data Unit project in which artificial intelligence solutions (such as text mining) are adopted to automatically extract both structured and unstructured data from hospital databases of patients infected from SARS- CoV-2. Feature selection and machine learning algorithms can be applied to develop diagnostic and prognostic support systems for clinicians.

The specific data that which will be exploited are:

* Demographics data;
* Patient comorbidities, vital signs and symptoms at the time of admission;
* Laboratory analysis;
* In-hospital complications (e.g.: need for non-invasive or invasive ventilation, access to intensive care unit, length of hospitalization, use of glucocorticoids or antibiotics, death);• Blood gas exchange information;
* Radiological reports;
* Medications at the time of admission, during hospitalization and at the time of discharge;
* Vaccination status.

Follow-up:

All patients will undergo a clinical follow-up by telephonic interview and/or clinical visit at 12 months from hospital discharge, during which the incidence of MACE, dysrhythmias, inflammatory heart disease and/or thrombotic disorders (both as incidence of the composite and as incidence of each individual components) in the past months will be investigate.

Primary endpoint:

To assess the presence of clinical predictors for the occurrence of myocardial injury, defined as at least one value of hs-cTnI >99th percentile upper reference limit (16), in patients hospitalized for COVID-19 infection.

Secondary endpoints:

1. The occurrence of myocardial injury during the index hospitalization for COVID-19 infection will be correlated with in-hospital complications (defined as the composite of the need for non-invasive or invasive ventilation, access to intensive care unit, length of hospitalization, use of glucocorticoids or antibiotics, and death).
2. The occurrence of myocardial injury in patients during the index hospitalization for COVID-19 infection will be included in a prediction model and correlated with future cardiovascular events (MACE), dysrhythmias, inflammatory heart disease and/or thrombotic disorders at 12-months follow-up.

Sample size calculation:

A comprehensive characterization of myocardial injury in COVID-19 infection is still lacking, and no clinical predictors of myocardial injury have been identified yet. Moreover, the long-term cardiovascular outcome of myocardial injury in the post-acute COVID-19 phase is largely unknown. Thus, this configures as a pilot study on large-scale cohort. As such no formal sample size calculation is needed. However, based on the COVID-19 datamart of our clinical institution and on inclusion criteria, the investigators expect to include in the study around 2000 patients hospitalized with COVID-19. Such a sample size is largely consistent with common rules of thumb for pilot studies. In addition, the estimated sample size is largely consistent with the van Smeden metamodels related to the new statistical approaches for the development of clinical prediction models (17). The square root of the mean squared prediction error (rMPSE) and mean absolute prediction error (MAPE) may be approximated via the results of these. Lower values for rMSPE and MAPE indicate better performance. For instance, at a sample size of N=400, with P=8 candidate predictors and an expected event fraction of 1⁄4, the predicted out-of-sample rMPSE would be 0.065 when ML model (without variable selection) is applied, and 0.053 for Ridge regression; MAPE would instead be 0.045 for the ML model and 0.038 for the Ridge regression.

Statistical analysis:

All demographic, clinical and laboratory characteristics will be summarized by descriptive statistics techniques. In depth, qualitative variables will be expressed by absolute and relative percentage frequencies. Quantitative variables, indeed, will be reported either as mean and standard deviation (SD) or median and interquartile range (IQR), respectively in the case they were normally or not normally distributed. Their distribution will be previously assessed by the Shapiro Wilk test. Between groups differences in the demographic, clinical, laboratory and pathologic features will be assessed by the Chi Square or the Fisher's exact test as for qualitative variables, with Yates correction, as appropriate,whilst quantitative variables will be evaluated either by the Student's t test or the Mann-Whitney U test, according to their distribution. Univariable and multivariable logistic regression models will be performed to evaluate the presence of clinical predictors for the occurrence of myocardial injury in COVID-19 infection. Results will be expressed as odds ratio (OR) with 95% confidence interval (CI). Model calibration performances will be evaluated via the Hosmer-Lemeshow goodness of fit test with 10 groups. Model performance will be assessed through receiver-operator characteristic (ROC) curve analysis by reporting the area under the curve, sensitivity, specificity and +/- likelihood ratio (LR).

Univariable and multivariable logistic regression analysis will be performed also to assess the association of myocardial injury in COVID-19 infection with in-hospital complications and need for aggressive therapies. Finally, to assess whether the presence of myocardial injury during COVID-19 predicts a worse outcome, in term of both MACEs at 12 months and single components, uni- and multivariable interaction proportional hazard Cox regression models will be computed. The investigators will consider, as for MACEs, time to first event, and for each component, time to each event.

To evaluate combined effects between each clinical/laboratory predictor and presence/absence of Myocardial Injury (MI), multivariable interaction Cox models will be fitted, and the interaction hazard ratios (IHR) evaluated. In particular, for each predictor, one interaction Cox model will be fitted. In this framework, IHR = 1 indicates no synergy between predictor and MI, IHR <1 expresses a reduction of hazard due to the synergy, while IHR >1 an increased hazard. The interaction parameters (IHR) will be interpreted as difference (in HR terms) of the predictor and MI (absence of MI as reference category).

Proportionality of the hazard functions will be assessed by visual inspection of hazard plots and Schoenfeld residuals. When proportionality was doubtful, weighted Cox regression models would be fitted.

A two-tailed analysis will be performed and a p value <0.05 will be considered as statistically significant. Statistical analyses will be performed using R software version 4.2.1 (CRAN ®, R Core 2021) (and its packages survival, survminer, coxphw and Hmisc) (18).

A pre-specified analysis to assess the preditors of myocardial injury across different age groups (< or = 60-year, 61-75-year, and > or = 75-year) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Overt COVID-19 infection (molecular nasopharyngeal swab positive for SARS-CoV-2 ≥1);
* Patient with at least a high sensitivity Troponin I measured during hospitalization course.
* Available data on vaccination.
* Verbal informed consent

Exclusion Criteria:

* Age <18 years;
* Patient in whom at least one high sensitivity Troponin I value measured during the course of hospitalization is not available.
* No data available on vaccination status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients hospitalized at Policlinico Universitario A. Gemelli IRCSS since March 1, 2021, with a diagnosis of SARS-CoV-2 infection (≥1 positive nasopharyngeal swab) and at least one value of high-sensitivity cardiac troponin I (hs-cTnI) measured during the index hospitalization will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
To identify the clinical predictors of myocardial injury | Up to 30 days
  Th occurence of clinical predictors of myocardial injury during the index hospitalization (defined as at least one value of hs-cTnI >99th percentile upper reference limit) will be evaluated using univariable and multivariable logistic regression models. Results will be expressed as odds ratio (OR) with 95% confidence interval (CI).

SECONDARY OUTCOMES:
To assess the correlation between myocardial injury and in-hospital complications | Up to 30 days
  The occurrence of myocardial injury during the index hospitalization for COVID-19 infection will be correlated with in-hospital complications (defined as the composite of the need for non-invasive or invasive ventilation, access to intensive care unit, length of hospitalization, use of glucocorticoids or antibiotics, and death) using univariable and multivariable logistic regression analysis.
To assess if myocardial injury can predict MACE at 1-year follow-up | 1 year
  The occurence of myocardial injury during the index hospitalization for COVID-19 infection will be included in a prediction model and correlated with MACE (defined as the composite of cardiovascular death, ischemic heart disease [acute or chronic coronary syndromes], stroke/transient ischemic attack [TIA] and hospitalization for heart failure), dysrhythmias, inflammatory heart disease and/or thrombotic disorders at 12-months follow-up using uni- and multivariable interaction proportional hazard Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco A Montone, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Li JW, Han TW, Woodward M, Anderson CS, Zhou H, Chen YD, Neal B. The impact of 2019 novel coronavirus on heart injury: A Systematic review and Meta-analysis. Prog Cardiovasc Dis. 2020 Jul-Aug;63(4):518-524. doi: 10.1016/j.pcad.2020.04.008. Epub 2020 Apr 16. PMID 32305557
- [Background] Bavishi C, Bonow RO, Trivedi V, Abbott JD, Messerli FH, Bhatt DL. Special Article - Acute myocardial injury in patients hospitalized with COVID-19 infection: A review. Prog Cardiovasc Dis. 2020 Sep-Oct;63(5):682-689. doi: 10.1016/j.pcad.2020.05.013. Epub 2020 Jun 6. PMID 32512122
- [Background] Al-Aly Z, Xie Y, Bowe B. High-dimensional characterization of post-acute sequelae of COVID-19. Nature. 2021 Jun;594(7862):259-264. doi: 10.1038/s41586-021-03553-9. Epub 2021 Apr 22. PMID 33887749
- [Background] Daugherty SE, Guo Y, Heath K, Dasmarinas MC, Jubilo KG, Samranvedhya J, Lipsitch M, Cohen K. Risk of clinical sequelae after the acute phase of SARS-CoV-2 infection: retrospective cohort study. BMJ. 2021 May 19;373:n1098. doi: 10.1136/bmj.n1098. PMID 34011492
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Xie Y, Xu E, Bowe B, Al-Aly Z. Long-term cardiovascular outcomes of COVID-19. Nat Med. 2022 Mar;28(3):583-590. doi: 10.1038/s41591-022-01689-3. Epub 2022 Feb 7. PMID 35132265
- [Background] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] van Smeden M, Moons KG, de Groot JA, Collins GS, Altman DG, Eijkemans MJ, Reitsma JB. Sample size for binary logistic prediction models: Beyond events per variable criteria. Stat Methods Med Res. 2019 Aug;28(8):2455-2474. doi: 10.1177/0962280218784726. Epub 2018 Jul 3. PMID 29966490

DOCUMENTS (1):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05392088/Prot_000.pdf